CLINICAL TRIAL: NCT05127967
Title: Phenotypic, Biological and Functional Consequences of Mutations in the SPG7 Gene at the Heterozygous State
Brief Title: Consequences of Mutations in the SPG7 Gene at the Heterozygous State
Acronym: CONSP-HET7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL20_0615
Record Dates: First submitted 2021-10-14; First posted 2021-11-19 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: SPG7
Keywords: SPG7; Dominant; human; Drosophila; mitochondria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with neurological symptoms and two mutations in the SPG7 gene (Other): Symptomatic patients with SPG7 mutations (homozygous or compound heterozygous)
  Interventions: Other: Skin biopsy
- Patients with neurological symptoms and one mutation in the SPG7 gene (Other): Patients presenting neurological symptoms corresponding to SPG7 disease (adult onset spastic ataxia with CPEO and/or optic atrophy) with only one mutation found in the SPG7 gene
  Interventions: Other: Skin biopsy
- Controls (Other): Patients without mutations in the SPG7 gene requiring spinal surgery because of a non-genetic neurologic disorders
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — A skin biopsy involves taking a piece of skin to obtain cells (fibroblasts). Skin biopsy is a minimally invasive examination and a technically simple procedure performed with a 3mm diameter punch, or with a scalpel under local anesthesia (Lidocaine patch). The procedure can be done in a consultation office with strict asepsis. It lasts 15 minutes in total + the time to reach between putting on the lidocaine patch and performing the procedure. This biopsy will usually be done on the inside of the arm. In the majority of cases, it is not helpful to close the scar with stitches.

SUMMARY:
Paraplegin, encoded by the SPG7 gene, is an ATP-dependent mAAA protease located in the inner mitochondrial membrane. Its function is not fully understood. Mutations in the SPG7 gene are responsible for spastic paraplegia type 7. Although spastic paraplegia type 7 is considered to be a recessive disease, some clinical observations also point to a detrimental effect of a variant in SPG7 in the heterozygous state. Thus, the presence of a single mutated variant of the SPG7 gene could be a risk factor for the development of neurological diseases. This has important implications for genetic counseling of patients and for the understanding of the function of the SPG7 protein and the mechanisms of disease development.

DETAILED DESCRIPTION:
Although spastic paraplegia type 7 is considered to be a recessive disease, some clinical observations also argue for a detrimental effect of a variant in SPG7 in the heterozygous state. Thus, the presence of a single mutated variant of the SPG7 gene could be a risk factor for the development of neurological diseases. This has important implications for genetic counseling of patients and for the understanding of the function of the SPG7 protein and the mechanisms of disease development. To date there have been no studies to specifically explore the pathogenic role of single heterozygous variants in the SPG7 gene.

The aim of this project is to fully characterize different models expressing single heterozygous SPG7 mutations in order to detect phenotypical, biological or functional alterations. In particular, the investigators will conduct analysis on fibroblasts from symptomatic patients with mutations in the SPG7 gene (homozygous, compound heterozygous or single heterozygous), and controls. Cellular models will be particularly useful in order to study an alteration in calcium homeostasis and in the response to ER stressors. In parallel, studies will be performed using the genetic animal model of Drosophila melanogaster.

ELIGIBILITY:
Case inclusion criteria

* age > or equal to 18 years
* presence of neurological symptoms compatible with GSP7 (ataxia, spasticity progressive external ophthalmoplegia, and/or optic atrophy)
* presence of two mutations in the SPG7 gene (= recessive forms of SPG7) or of a single mutation in the simple heterozygous state in the absence of other genetic factors explaining the symptoms

Inclusion criteria for controls

* Age > or equal to 18 years
* Subject who is already undergoing neurosurgical intervention as part of the care pathway for an for an acquired, non-genetic neurological problem (e.g. herniated disc, narrow lumbar canal)

Non-inclusion Criteria of cases

* Refusal to sign the written informed consent signed by the patient (or by his representative in case of a patient under guardianship.
* Patients with specific contraindications for skin biopsy current anticoagulant treatment; any pathologies that may cause a risk of bleeding (e.g. hemophiliacs)
* Refusal of the patient, of the guardian if necessary, to sign the informed consent to participate in the in the research
* Not being a beneficiary of a social protection plan Patient deprived of liberty

Non-inclusion Criteria of controls

* Patients with a genetic neurological disease or mitochondrial disease
* Patients with specific contraindications for skin biopsy: current anticoagulant treatment; all pathologies that may cause a risk of bleeding (e.g. hemophilia)
* Refusal to sign the informed consent to participate in the research
* Not benefiting from a social protection plan
* Patient deprived of liberty
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiratory activity measured by Seahorse analyser and quantification of mADN vs nuclear AND in activity in patients with neurological symptoms and one or two mutations in the SPG7 gene vs controls | Inclusion
Mitochondrial dimension and morphology by electronic microscopy and quantification of mitochondrial motility by direct imaging activity in patients with neurological symptoms and one or two mutations in the SPG7 gene vs controls | Inclusion

SECONDARY OUTCOMES:
Mitochondrial calcium quantification after expression of a probe for calcium detection in patients with neurological symptoms and one or two mutations in the SPG7 gene vs controls | Inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, Herault, France